CLINICAL TRIAL: NCT05589636
Title: A Randomized Controlled Intervention Study to Assess the Effect of Bergamot Juice on LDL Cholesterol Level in Healthy Subjects
Brief Title: Effect of Bergamot Juice on LDL Cholesterol Level in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Collaborators: University of Parma (Other)
Responsible Party: Principal Investigator, Alessandra Dei Cas, Associate Professor, University of Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 562/2021/SPER /UNIPR
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bergamot juice (Experimental): Consumption of 400 cc/die of Bergamot juice (35% in water sweetened with stevia) for 12 weeks
  Interventions: Dietary Supplement: Bergamot Juice
- Free diet (No Intervention): Free diet

INTERVENTIONS:
Dietary Supplement: Bergamot Juice — Bergamot Juice (35% in water)
  Arms: Bergamot juice

SUMMARY:
A single-centre, randomized (1:1), open label, controlled study to assess the lipid-lowering effect at 12 weeks of 400 cc/die bergamot juice consumption compared to free diet in healthy subjects

DETAILED DESCRIPTION:
Cardiovascular diseases (CV) are the first cause of morbidity and mortality in industrialized countries. Hypercholesterolemia is the main CV risk factor: high cholesterol values are directly and linearly correlated with CV events and mortality in the absence of a threshold value. Intervention studies show unequivocally how the decrease in cholesterol levels significantly reduces CV risk. Bergamot juice is considered a possible food with nutraceutical activity, especially as regards the control of blood cholesterol levels. It is now known that bergamot juice has chemical components that can positively affect blood cholesterol levels. These compounds are called 3-hydroxy-3-methyl flavonoids (HMG-flavonoids) and are peculiar to some citrus plants and in particular to the Citrus bergamia species. The aim of this study is to provide clinical evidence of the effect of these metabolites on cholesterol levels. Specifically, a single-centre, randomized (1:1), open label, controlled study is conducted in healthy subjects to evaluate the possible lipid-lowering effects at 12 weeks of 400 cc/die of bergamot juice consumption compared to a free diet. Changes in the following parameters: body mass index (BMI kg/m²), waist circumference, glycemia, insulin, glycated hemoglobin (HbA1C), total cholesterol, HDL cholesterol and triglycerides, plasma levels of inflammatory cytokines, C-reactive protein (hsCRP) and Proprotein convertase subtilisin / kexin type 9 (PCSK9) are also investigated at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian persons of both sexes aged ≥18 and ≤75 years
* ability to understand the methods, purposes and implications of the study, and to give free and informed consent

Exclusion Criteria:

* Diabetes mellitus defined according to ADA criteria
* Present or past history of alcohol or drug abuse or organ failure (kidney and liver)
* Tumor pathologies in the last 5 years;
* Past or present cerebro-vascular diseases;
* Subjects taking drugs or supplements active on the lipid profile;
* Pregnancy or breastfeeding
* Presence of severe or monogenic dyslipidemia
* Use of antibiotics in the last three months before enrollment
* Subjects who are on a diet for any reason
* Individuals who have intentionally or unintentionally lost 3 kg or more of body weight in the past 3 months.
* Known allergies to some components of the product
* Subjects who do not like bergamot

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Low-density lipoprotein (LDL) cholesterol | 12 weeks
  Changes in LDL cholesterol at 12 weeks in both study arms

SECONDARY OUTCOMES:
body mass index (BMI) | 12 weeks
  Changes in body mass index (BMI) at 12 weeks in both study arms
waist circumference | 12 weeks
  Changes in waist circumference at 12 weeks in both study arms
fasting plasma glucose (FPG) | 12 weeks
  Changes in FPG at 12 weeks in both study arms
insulinemia | 12 weeks
  Changes in insulinemia at 12 weeks in both study arms
glycated hemoglobin | 12 weeks
  Changes in glycated hemoglobin at 12 weeks in both study arms
total cholesterol | 12 weeks
  Changes in total cholesterol at 12 weeks in both study arms
high density lipoprotein (HDL) cholesterol | 12 weeks
  Changes in HDL cholesterol at 12 weeks in both study arms
triglycerides | 12 weeks
  Changes in triglycerides at 12 weeks in both study arms
plasma levels of inflammatory cytokines | 12 weeks
  Changes in plasma levels of inflammatory cytokines (IL-1,IL-6,IL-10,hsPCR,TNF-alpha) at 12 weeks in both study arms
Proprotein convertase subtilisin/kexin type 9 (PCSK9) | 12 weeks
  Changes in PCSK9 at 12 weeks in both study arms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Parma, Department of Medicine and Surgery, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballistreri G, Amenta M, Fabroni S, Consoli V, Grosso S, Vanella L, Sorrenti V, Rapisarda P. Evaluation of lipid and cholesterol-lowering effect of bioflavonoids from bergamot extract. Nat Prod Res. 2021 Dec;35(23):5378-5383. doi: 10.1080/14786419.2020.1768085. Epub 2020 May 22. PMID 32441543
- [Background] Cappello AR, Dolce V, Iacopetta D, Martello M, Fiorillo M, Curcio R, Muto L, Dhanyalayam D. Bergamot (Citrus bergamia Risso) Flavonoids and Their Potential Benefits in Human Hyperlipidemia and Atherosclerosis: an Overview. Mini Rev Med Chem. 2016;16(8):619-29. doi: 10.2174/1389557515666150709110222. PMID 26156545
- [Background] Di Donna L, De Luca G, Mazzotti F, Napoli A, Salerno R, Taverna D, Sindona G. Statin-like principles of bergamot fruit (Citrus bergamia): isolation of 3-hydroxymethylglutaryl flavonoid glycosides. J Nat Prod. 2009 Jul;72(7):1352-4. doi: 10.1021/np900096w. PMID 19572741
- [Background] Ference BA, Ginsberg HN, Graham I, Ray KK, Packard CJ, Bruckert E, Hegele RA, Krauss RM, Raal FJ, Schunkert H, Watts GF, Boren J, Fazio S, Horton JD, Masana L, Nicholls SJ, Nordestgaard BG, van de Sluis B, Taskinen MR, Tokgozoglu L, Landmesser U, Laufs U, Wiklund O, Stock JK, Chapman MJ, Catapano AL. Low-density lipoproteins cause atherosclerotic cardiovascular disease. 1. Evidence from genetic, epidemiologic, and clinical studies. A consensus statement from the European Atherosclerosis Society Consensus Panel. Eur Heart J. 2017 Aug 21;38(32):2459-2472. doi: 10.1093/eurheartj/ehx144. PMID 28444290
- [Background] Silverman MG, Ference BA, Im K, Wiviott SD, Giugliano RP, Grundy SM, Braunwald E, Sabatine MS. Association Between Lowering LDL-C and Cardiovascular Risk Reduction Among Different Therapeutic Interventions: A Systematic Review and Meta-analysis. JAMA. 2016 Sep 27;316(12):1289-97. doi: 10.1001/jama.2016.13985. PMID 27673306